CLINICAL TRIAL: NCT05717049
Title: Theophylline Effects in the Fontan Circulation (THIEF Pilot Study)
Brief Title: Theophylline Effects in the Fontan Circulation
Acronym: THIEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Norwegian Health Association (Other); Norwegian Association for Children with Congenital Heart Disease (Unknown)
Responsible Party: Principal Investigator, Thomas Möller, Principal investigator, MD PhD, senior consultant / senior researcher, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU CT 2022-500301-41-00
Record Dates: First submitted 2023-01-16; First posted 2023-02-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Congenital Heart Disease
Keywords: Fontan circulation; Cardiorespiratory fitness; Pulmonary function; Cardiac function; Quality of life
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): 12 week oral treatment (theophylline)
  Interventions: Drug: Theophylline Tablets

INTERVENTIONS:
Drug: Theophylline Tablets — 12 week oral treatment
  Other Names: ATC R03D A04

SUMMARY:
A single group treatment phase 2 single-arm no-masking study to assess safety and efficacy of a short-term oral treatment with theophylline (ATC-no. R03D A04) in terms of improvements in cardiorespiratory fitness, health-related quality of life, cardiac performance and respiratory function in male and female adolescents aged 16 to 25 years with a Fontan-type surgical palliation of univentricular congenital heart disease.

DETAILED DESCRIPTION:
Single-group uncontrolled single-center open-label treatment study in adolescents (age 16-25 years) with univentricular congenital heart defects surgically palliated with a Fontan-type operation. Inclusion of eligible patients from inpatient and outpatient contacts at participating departments at Oslo University Hospital Rikshospitalet.

Study inclusion visit, drug treatment, remote dose adjustment, heart rhythm monitoring, and final post-treatment assessment study visit will be performed at the clinical research ward for children, Division of Paediatric and Adolescent Medicine.

Dose adjustment decisions and heart rhythm monitoring will be effectuated by the medical monitors (pediatric cardiology, cardiology) with continuous service through the entire study period.

Study duration: approximately 6 months (depending on inclusion progress, from inclusion of first participant until final visit of last enrolled participant) Individual treatment duration: minimum 12 weeks, maximum 15 weeks or until final study visit.

Visit frequency: two study visits, at inclusion and at end of treatment period (earliest after 12 weeks of treatment and latest after 15 weeks of treatment).

Number of Participants: Ten participants with both genders represented will be enrolled and invited to the study inclusion visit to achieve an intervention group of 10 individuals starting the oral treatment. In terms of being a pilot study, the study will also help to estimate the expected fractions of evaluable and non-evaluable participant in a subsequent full scale randomized clinical trial. Evaluability means the participant absolving all included study tests during inclusion and final study visit and completing scheduled dosage control and ECG monitoring tasks.

Health measurement / observation:

At inclusion and final visit:

* Demographics, biometric data, medical history
* Quality of life assessment by questionnaire (SF-36, EQ-5D)
* Echocardiography for cardiac function assessment
* Pulmonary function test incl. diffusion capacity
* Cardiopulmonary exercise test (bicycle ergometer)
* Home-based polysomnography

During treatment phase:

* Dosage monitoring by analysis of theophylline concentration in blood sample (obtained locally) in addition to analysis of liver and renal parameters (ALT, bilirubin, creatinine), repeated on indication (after dose adjustment, in case of arrhythmic events)
* Treatment compliance and AE monitoring by symptom report in electronic participant log book in ViedocMe (part of the eCRF-database)
* ECG-monitoring (rhythm storage at least every hour) by tape-on ECG-device (ECG247®) connected to via smartphone app to an online database with 24/7 accessibility for medical monitor (1).

During early intervention phase until 5-7 days after therapeutic drug concentration is achieved, the participant will continuously use the ECG247 device. In case of symptoms (palpitations or other arrhythmia-suspect symptoms), the participant will be able to notify the medical monitor (cardiologist) for immediate review of ECG readings. After cessation of continuous ECG-monitoring, the participant will be equipped with additional ECG-tapes for symptom-initiated ECG-readings and contact with medical monitor as needed.

Drug regimen / adjustments:

After inclusion visit, the participant starts on oral study medication (theophylline depot tablets 200mg, start dose 200mg bid).

After 3-5 days, the participant visits the family physician or a nearby hospital laboratory to collect a blood sample 4-6 hours after drug intake which is shipped to OUS for analysis (serum concentration of theophylline, creatinine, ALAT, bilirubin). Target concentration of theophylline during study period is 30-80 μmol/Liter. Dose adjustments, if needed, are made by a physician at the research unit in collaboration with the PI. Dose increase or decrease depending on serum concentration and drug tolerance by 100mg steps up or down, i.e., from 200mg bid to either 100mg bid or 300mg bid (see also algorithm in section 6.5 Dose Modification). Any dosing change has to be followed by repeat blood work after 3-5 days and renewed review of theophylline concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with univentricular congenital heart disease with a Fontan-type palliation

   1. Who are able to perform all diagnostic and monitoring procedures necessary during trial period, in particular being able to perform a symptom-limited cardiopulmonary exercise test on an upright ergometer bicycle.
   2. With available hepatic imaging results (ultrasound or magnetic resonance imaging) from less than 12 months before inclusion
   3. Without biochemical indications of more than mild liver disease or liver failure (se exclusion criteria) of more than mildly reduced kidney function.
   4. Considered and assessed eligible for administration of Theo-Dur® (theophylline) as specified in the SmPC.
2. Body mass index (BMI) within the range 18.5 - 34.9 kg/m2 (inclusive).
3. Contraceptive use by women is not under any national / local regulations in Norway.

   1. Male participants: no restrictions.
   2. Female participants: female participants should have a negative pregnancy test at inclusion and they receive information prior to consent that onset of pregnancy during treatment period has to be reported to the study team and leads to exclusion.
4. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

For participants < 18 years, all (both) parents or caregivers with parental responsibilities have to sign the consent form in addition to the participant.

Exclusion Criteria:

1. Current or previous (last 12 months) tachyarrhythmia which has been cause of medical investigation or hospitalization.
2. Heart rhythm during inclusion visit other than:

   * sinus rhythm or regular supraventricular rhythm (visible P-waves) regardless P-wave angle
   * nodal rhythm
   * isolated extra beats (supraventricular or ventricular) of a frequency considered clinically non-significant
3. Systemic hypertension (systolic or diastolic blood pressure above 95 percentile)
4. Biochemical signs of more than mild liver disease or liver failure indicated by one of the following:

   1. INR > 1.5 in the absence of warfarin treatment,
   2. ALAT more than twice the upper normal limit
   3. Bilirubin more than twice the upper normal limit
5. Imaging signs from the recent 12 months indicating more than mild Fontan-associated liver disease, indicated by imaging findings that need further diagnostic work-up to rule out hepato-cellular carcinoma
6. Biochemical indication of more than mildly reduced kidney function indicated by:

   a. Creatinine > 150 μmol/L (male) or > 120 μmol/L (female)
7. Pregnancy
8. Inherited forms of galactose intolerance (Lapp lactase deficiency or glucose-galactose malabsorption
9. Hypersensitivity to theophylline
10. Current treatment with pulmonary vasodilator medication (sildenafil, tadalafil, udenafil, bosentan, ambrisentan, macicentan, or any prostacyclin derivate)
11. Ongoing pharmacological treatment with the risk of drug-drug interactions. (Examples: cimetidine, quinolone derivates like enoxacin, ciprofloxacin, perfloxacin, viloxazine, macrolide antibiotics like erythromycin, troleandomycin, allopurinol, propranolol, disulfiram, isoniazid, oral contraceptives, flu vaccine, mexiletine, nifedipine, norfloxacin, ranitidin, tiabendazol, verapamil, fluvoxamine, carbamazepine, felodipine, phenobarbital, phenytoin, rifampicin, lithium, ketamine, glucagon)
12. Pregnancy or breastfeeding

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety - adverse events | 12 weeks
  Frequency of treatment emerged AE/SAE
Feasibility and safety - tolerability | 12 weeks
  Freedom from participant dropout based on tolerability of the study intervention
Feasibility and safety - drug dosing | 12 weeks
  Number of participants requiring dose reduction after first serum concentration
Feasibility and safety - arrhythmia | 12 weeks
  Freedom of arrhythmogenic side effects of the study treatment leading to patient dropout
Cardiorespiratory fitness | 12 weeks
  Difference in oxygen uptake at anaerobic/ventilatory threshold pre/post treatment

SECONDARY OUTCOMES:
Health-related quality-of-life | 12 weeks
  Difference inn total scores from EQ-5D-5L questionnaires pre/post treatment (single digit score (0-5 = "no problems" to "extreme problems") for five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression))
Health-related quality-of-life (SF 36) | 12 weeks
  Difference inn total scores from SF-36 questionnaire pre/post treatment (36 items scored scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100 respectively)
Cardiac performance | 12 weeks
  Ventricular function as assessed by echocardiography at rest pre/post treatment
Respiratory function | 12 weeks
  Diffusion capacity pre/post treatment
Sleep disordered breathing | 12 weeks
  Change in Apnea Hypopnea Index during home-based sleep study pre-/post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Möller, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Department of Paediatric Cardiology, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EU Clinical Trials database, use search term "theophylline" — https://euclinicaltrials.eu/search-for-clinical-trials/

DOCUMENTS (1):
  • Study Protocol (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT05717049/Prot_001.pdf